CLINICAL TRIAL: NCT06891157
Title: Chidamide Plus R-CHOP (CR-CHOP) in Newly Diagnosed Double-Expressor Diffuse Large B-Cell Lymphoma With Other Molecular Subtypes: A Prospective, Multicenter Phase II Trial
Brief Title: Chidamide Plus R-CHOP in Newly Diagnosed Double-Expressor Diffuse Large B-Cell Lymphoma With Other Molecular Subtypes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-1157
Record Dates: First submitted 2025-03-13; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chidamide; R-CHOP Chemotherapy; DLBCL - Diffuse Large B Cell Lymphoma; Double-expressor Lymphoma (DEL)
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CR-CHOP arm (Experimental): Newly Diagnosed DEL Patients Receiving Chidamide plus R-CHOP(Rituximab、Cyclophosphamide、Doxorubicin、Vincristine and Prednisone) Regimen Treatment
  Interventions: Drug: Chidamide plus R-CHOP

INTERVENTIONS:
Drug: Chidamide plus R-CHOP — Chidamide Plus R-CHOP (Rituximab、Cyclophosphamide、Doxorubicin、Vincristine and Prednisone)

SUMMARY:
Evaluation of the Safety and Efficacy of CR-CHOP Treatment in Newly Diagnosed Double-Expressor DLBCL with Other Molecular Subtypes

DETAILED DESCRIPTION:
Patients with the Other Molecular Subtype of double-expressor diffuse large B-cell lymphoma (DEL-DLBCL) demonstrate significantly poorer survival outcomes. The DEB trial demonstrated that chidamide combined with R-CHOP significantly improves the complete response (CR) rate in DEL patients and shows a definitive trend toward benefit in event-free survival (EFS). Therefore, we plan to evaluate the efficacy and safety of C-R-CHOP (chidamide plus R-CHOP) in treating DLBCL patients with the DEL Other molecular subtype.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for enrollment:

  1. ≥18 years of age;
  2. Diffuse large B-cell lymphoma diagnosed by pathological diagnosis according to WHO 2016 classification criteria;
  3. Molecular subtyping, determined through high-throughput sequencing of pathological tissue or peripheral blood, is categorized as the "Other" subtype;
  4. Immunohistochemistry revealed overexpression of MYC and BCL2: MYC ≥ 40%, BCL2 ≥ 50%;
  5. Measurable lesions identified on cross-sectional imaging through diagnostic modalities (computed tomography [CT] or magnetic resonance imaging [MRI]) are defined as the presence of at least one two-dimensional lesion with a maximum cross-sectional diameter (GTD) ≥1.5 cm, irrespective of the short-axis diameter;
  6. The Eastern Cooperative Oncology Group (ECOG) performance status score is ≤2；
  7. Adequate hepatic function is defined as: total bilirubin (TBIL) ≤ 3 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5 × ULN; alkaline phosphatase (ALP) ≤ 5 × ULN; serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 35 mL/min as calculated by the Cockcroft-Gault formula;
  8. Voluntary participation with willingness to provide the aforementioned treatment data, accompanied by a signed and dated informed consent form.

     Exclusion Criteria:
* Patients who meet any of the following criteria will be excluded from the study：

  1. Currently enrolled in another clinical trial；
  2. Received prior lymphoma treatment with alternative regimens before enrollment;
  3. Presence of concurrent malignant tumors;
  4. Deemed ineligible for participation by the investigator's judgment；
  5. Presence of severe psychiatric or neurological disorders that may impair the ability to provide informed consent and/or affect the reporting or observation of adverse events；
  6. Patients unable to comply with follow-up requirements；
  7. Pregnant or lactating women, and patients of childbearing potential unwilling to use contraception;
  8. Active infection or uncontrolled HBV (HBsAg positive and/or HBcAb positive and HBV DNA positive), HCV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2027-08-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  from date of inclusion to date of progression, relapse, or death from any cause

SECONDARY OUTCOMES:
CR rate | up to 6 cycles (each cycle is 21 days)
  complete remission rate
OS | 2 years
  Overall Survival: from the date of inclusion to date of death, irrespective of cause
ORR | up to 6 cycles (each cycle is 21 days)
  The Overall Response Rate

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China